CLINICAL TRIAL: NCT02083107
Title: COMPARISON BETWEEN RECTAL & SUBLINGUAL MISOPROSTOL BEFORE CAESARIAN SECTION TO REDUCE INTRA & POST-OPERATIVE BLOOD LOSS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Mohamed S. Sweed, Lecturer of Obstetrics &Gynecology, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 9021344
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-11

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum hemorrhage; Intrapartum blood loss; Misoprostol
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sublingual misoprostol & rectal placebo (Experimental): will receive 400 microgram of misoprostol (Sigma) sublingual "2 tablets" and rectal placebo"2 tablets".
  Interventions: Drug: Misoprostol
- rectal & sublingual placebo (Placebo Comparator): will receive rectal placebo"2 tablets" and sublingual placebo"2 tablets".
  Interventions: Other: Placebo
- rectal misoprostol & sublingual placebo (Experimental): will receive 400 microgram of misoprostol (Sigma) rectal "2 tablets" and sublingual placebo"2 tablets".
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Comparison of different routes of administration of 400 micro gram misoprostol
  Other Names: Misotac; Cytotec
  Arms: rectal misoprostol & sublingual placebo; sublingual misoprostol & rectal placebo
Other: Placebo
  Arms: rectal & sublingual placebo

SUMMARY:
The aim of the work is to evaluate & compare the effectiveness of rectally administered PGE1 synthetic analogue (misoprostol) 400 microgram versus sublingually administered misoprostol before caesarean section to decrease blood loss during and after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients booked for elective cesarean section.
2. Singleton pregnancies. 3- Full term pregnancies (GA 37-42 weeks). 4- Patients with only previous one cesarian section

Exclusion Criteria:

1. Primigravida.
2. Blood dyscrasias.
3. Large fibroids.
4. Multiple pregnancies.
5. Overdistended uterus eg. Hydramnios.
6. Pre-eclampsia.
7. Marked maternal anemia (Preoperative hemoglobin < 9 gm/dl).
8. Previous history of PPH.
9. Contraindications to prostaglandin therapy (e.g. history of severe bronchial asthma or allergy to misoprostol.
10. Placenta previa.
11. Contraindication to spinal anesthesia.
12. Previous myomectomy.
13. Previous two or more C.S.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 636 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S. Sweed, MD, Principal Investigator — Ain Shams University; Mourad M. El-Said, Professor, Study Director — AinShams University; Amgad E. Abou-Gamrah, Ass.Prof., Study Director — AinShams university; Haitham El-Sabe, MD, Study Director — AinShams University; Mohamed M. AbdEl-Hamid, Registrar, Principal Investigator — AinShams University
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sublingual Misoprostol & Rectal Placebo | Rectal & Sublingual Placebo | Rectal Misoprostol & Sublingual Placebo
Started | 212 (212 women received 2 tablets of Misotac® sublingually and 2 placebo tablets rectally.) | 212 (212 women received 2 tablets of placebo sublingually and 2 placebo tablets rectally.) | 212 (212 women received 2 tablets of Misotac® rectally and 2 placebo tablets sublingually.)
Completed | 212 (212 women received 2 tablets of Misotac® sublingually and 2 placebo tablets rectally.) | 212 (212 women received 2 tablets of placebo sublingually and 2 placebo tablets rectally.) | 212 (212 women received 2 tablets of Misotac® rectally and 2 placebo tablets sublingually.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sublingual Misoprostol & Rectal Placebo | Rectal & Sublingual Placebo | Rectal Misoprostol & Sublingual Placebo | Total
Number analyzed (Participants) | 212 | 212 | 212 | 636
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (2.6) | 26.4 (2.7) | 26.5 (2.5) | 26.6 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 212 | 212 | 636
  Male | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m2] | 27.5 (1.7) | 27.6 (1.9) | 27.4 (1.7) | 27.5 (1.76)
Parity [Median (Inter-Quartile Range); unit: Births] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
Gestational Age [Mean (Standard Deviation); unit: Weeks] | 38.9 (1) | 38.9 (0.9) | 38.8 (0.9) | 38.8 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Blood Loss
Time Frame: from start of cesarean section till the end of operation (average one hour)
Measure: Mean (Standard Deviation); unit: millilitres
Arm/Group | Sublingual Misoprostol & Rectal Placebo | Rectal & Sublingual Placebo | Rectal Misoprostol & Sublingual Placebo
Number analyzed (Participants) | 212 | 212 | 212
millilitres | 357.8 (129.7) | 641.7 (135.7) | 457.5 (140.7)

2. Secondary Outcome: Need for Extra Ecbolics (Oxytocin).
Time Frame: from start of cesarean section till the end of operation (average one hour)
Measure: Number; unit: participants
Arm/Group | Sublingual Misoprostol & Rectal Placebo | Rectal & Sublingual Placebo | Rectal Misoprostol & Sublingual Placebo
Number analyzed (Participants) | 212 | 212 | 212
participants | 209 | 206 | 204

3. Other Pre Specified Outcome: Change in Hemoglobin Concentration
Time Frame: 24 hours postoperative from baseline hemoglobin
Measure: Mean (Standard Deviation); unit: gram/dL
Arm/Group | Sublingual Misoprostol & Rectal Placebo | Rectal & Sublingual Placebo | Rectal Misoprostol & Sublingual Placebo
Number analyzed (Participants) | 212 | 212 | 212
gram/dL | -0.3 (0.1) | -0.9 (0.1) | -0.4 (0.1)

4. Secondary Outcome: APGAR Score
Description: The Apgar score is the first test given to a newborn, it is referred to as an acronym for: Appearance, Pulse, Grimace, Activity, and Respiration. Scores obtainable are between 10 and 0, with 10 being the highest possible score. Pulse: above 100 beats per minute (2), below 100 beats per minute (1), absent (0). Respiration: Normal rate and effort, good cry (2), Slow or irregular,weak cry (1), absent (0). Grimace: Pulls away, sneezes, coughs, or cries with stimulation (2), Facial movement only (1), absent (0). Activity: Active, spontaneous movement (2), Arms and legs flexed with little movement (1), absent (0). Appearance: Normal color (2), Normal color (but hands and feet are bluish) (1), Bluish-gray or pale all over (0).
Time Frame: 1minute and 5 minutes from delivery of the fetus
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sublingual Misoprostol & Rectal Placebo | Rectal & Sublingual Placebo | Rectal Misoprostol & Sublingual Placebo
Number analyzed (Participants) | 212 | 212 | 212
units on a scale
  APGAR 1 minute | 6.5 (0.5) | 6.5 (0.5) | 6.5 (0.5)
  APGAR 5 minute | 8.5 (0.5) | 8.5 (0.5) | 8.5 (0.5)

5. Secondary Outcome: Time to Resume Bowel Habits
Time Frame: average 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sublingual Misoprostol & Rectal Placebo | Rectal & Sublingual Placebo | Rectal Misoprostol & Sublingual Placebo
Number analyzed (Participants) | 212 | 212 | 212
hours | 15.1 (3.1) | 14.7 (3.5) | 14.5 (3.5)

6. Secondary Outcome: Need for Extra Analgesics
Time Frame: average 24 hours
Measure: Number; unit: participants
Arm/Group | Sublingual Misoprostol & Rectal Placebo | Rectal & Sublingual Placebo | Rectal Misoprostol & Sublingual Placebo
Number analyzed (Participants) | 212 | 212 | 212
participants | 56 | 62 | 50

7. Secondary Outcome: Need for Postoperative Blood Transfusion
Time Frame: average 24 hours
Measure: Number; unit: participants
Arm/Group | Sublingual Misoprostol & Rectal Placebo | Rectal & Sublingual Placebo | Rectal Misoprostol & Sublingual Placebo
Number analyzed (Participants) | 212 | 212 | 212
participants | 4 | 10 | 5

8. Secondary Outcome: Incidence of Wound Sepsis
Time Frame: upto one week
Measure: Number; unit: no. of cases experiencing wound sepsis
Arm/Group | Sublingual Misoprostol & Rectal Placebo | Rectal & Sublingual Placebo | Rectal Misoprostol & Sublingual Placebo
Number analyzed (Participants) | 212 | 212 | 212
no. of cases experiencing wound sepsis | 3 | 5 | 4

9. Secondary Outcome: Incidence of Adverse Effects
Time Frame: 24 hours
Measure: Number; unit: no. of cases experiencing side effects
Arm/Group | Sublingual Misoprostol & Rectal Placebo | Rectal & Sublingual Placebo | Rectal Misoprostol & Sublingual Placebo
Number analyzed (Participants) | 212 | 212 | 212
no. of cases experiencing side effects
  Fever | 44 | 11 | 26
  Chills | 42 | 11 | 24

10. Other Pre Specified Outcome: Change in Hematocrite Value
Time Frame: 24 hours postoperative from baseline hematocrite value
Measure: Mean (Standard Deviation); unit: Percentage Hematocrit
Arm/Group | Sublingual Misoprostol & Rectal Placebo | Rectal & Sublingual Placebo | Rectal Misoprostol & Sublingual Placebo
Number analyzed (Participants) | 212 | 212 | 212
Percentage Hematocrit | -0.1 (0.8) | -1.6 (0.3) | -0.1 (0.9)

ADVERSE EVENTS:
Time Frame: starting intra-operative till one week postoperative (time of checking the wound)
Arm/Group | Sublingual Misoprostol & Rectal Placebo | Rectal & Sublingual Placebo | Rectal Misoprostol & Sublingual Placebo
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/212 | 0/212
Other Adverse Events (participants affected / at risk) | 44/212 | 11/212 | 26/212
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sublingual Misoprostol & Rectal Placebo (N=212) | Rectal & Sublingual Placebo (N=212) | Rectal Misoprostol & Sublingual Placebo (N=212)
Fever (General disorders) | 44 | 11 | 26
wound sepsis (Infections and infestations) | 3 | 5 | 4
Chills (General disorders) | 42 | 11 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes